CLINICAL TRIAL: NCT00548860
Title: A Multi-center, Randomized Controlled Study to Investigate the Safety and Tolerability of IV Ferric Carboxymaltose (FCM) vs Standard of Care in Treating Iron Deficiency Anemia in Heavy Uterine Bleeding and Post Partum Patients
Brief Title: Safety of FCM vs. Standard of Care in Treating Iron Deficiency Anemia in Heavy Uterine Bleeding and Post Partum Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: American Regent, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1VIT07017
Record Dates: First submitted 2007-10-22; First posted 2007-10-24 (Estimated); Results first posted 2015-05-29 (Estimated); Last update posted 2018-02-20 (Actual); Status verified 2018-01

CONDITIONS: Anemia
MeSH Terms: conditions — Anemia | interventions — ferric carboxymaltose

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ferric Carboxymaltose (FCM) (Experimental): Undiluted dose of iron as FCM IV (15 mg/kg up to a maximum of 1000 mg)
  Interventions: Drug: Ferric Carboxymaltose
- Standard Medical Care (SMC) (Active Comparator): Varied as determined by the Investigator
  Interventions: Drug: Standard Medical Care (SMC)

INTERVENTIONS:
Drug: Ferric Carboxymaltose
  Arms: Ferric Carboxymaltose (FCM)
Drug: Standard Medical Care (SMC)
  Arms: Standard Medical Care (SMC)

SUMMARY:
The Objective of this study is to study the safety of FCM in patients with anemia caused by Heavy Uterine Bleeding and the Post Partum state.

ELIGIBILITY:
Inclusion Criteria:

* Female with iron deficiency anemia
* Hg </= 11 g/dL

Exclusion Criteria:

* Previous participation in a FCM trial
* Known Hypersensitivity to FCM
* History of anemia other that anemia due to heavy uterine bleeding or the post partum state
* current history of GI bleeding
* Received IV Iron within the month prior
* Anticipated need for surgery
* Malignancy history
* AST or ALT greater than normal
* Received an investigational drug within 30 days of screening
* Pregnant or sexually active females who are not willing ot use an effective form of birth control

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2018 (Actual)
Dates: Start 2007-10; Primary Completion 2009-03 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Luitpold Pharmaceuticals, Norristown, Pennsylvania, United States

REFERENCES:
- [Derived] Seid MH, Butcher AD, Chatwani A. Ferric Carboxymaltose as Treatment in Women with Iron-Deficiency Anemia. Anemia. 2017;2017:9642027. doi: 10.1155/2017/9642027. Epub 2017 Apr 13. PMID 28487769

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Hospitals and medical clinics
Groups:
- Ferric Carboxymaltose (FCM): Intravenous (IV) iron
- Standard Medical Care (SMC): SMC for postpartum and heavy uterine bleeding subjects with anemia
Period: Overall Study
Arm/Group | Ferric Carboxymaltose (FCM) | Standard Medical Care (SMC)
Started | 996 | 1022
Completed | 860 | 847
Not Completed | 136 | 175

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ferric Carboxymaltose (FCM) | Standard Medical Care (SMC) | Total
Number analyzed (Participants) | 996 | 1022 | 2018
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 25 | 27 | 52
  Between 18 and 65 years | 971 | 995 | 1966
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.2 (9.36) | 31.4 (8.98) | 31.3 (9.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 996 | 1022 | 2018
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 996 | 1022 | 2018

OUTCOME MEASURES:

1. Primary Outcome: Evaluate the Safety of the Maximum Administered Dose, 15 mg/kg (up to a Maximum 1,000 mg) of FCM Compared to SMC.
Description: Evaluate the safety of the maximum administered dose, 15 mg/kg (up to a maximum 1,000 mg) of FCM compared to SMC. The primary safety endpoint was the incidence of Serious Adverse Events (SAE's).
Time Frame: From Day 0 through 30 days after the last dose of study drug.
Measure: Number; unit: participants
Arm/Group | Ferric Carboxymaltose (FCM) | Standard Medical Care (SMC)
Number analyzed (Participants) | 996 | 1022
participants | 6 | 22

ADVERSE EVENTS:
Time Frame: 1 year and 5 months
Arm/Group | Ferric Carboxymaltose (FCM) | Standard Medical Care (SMC)
Serious Adverse Events (participants affected / at risk) | 6/996 | 22/1022
Other Adverse Events (participants affected / at risk) | 9/996 | 79/1022
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ferric Carboxymaltose (FCM) (N=996) | Standard Medical Care (SMC) (N=1022)
Anemia (Blood and lymphatic system disorders) | 1 | 0
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 1
Abdominal adhesions (Gastrointestinal disorders) | 0 | 1
Abdominal hernia (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 1
Necrotising Fasciitis (Infections and infestations) | 1 | 0
Postoperative abscess (Infections and infestations) | 1 | 0
Endometritis (Infections and infestations) | 0 | 1
Pyelonephritis (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Postpartum hemorrhage (Pregnancy, puerperium and perinatal conditions) | 0 | 2
Retained placenta or membranes (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Uterine hemorrhage (Reproductive system and breast disorders) | 1 | 5
Menorrhagia (Reproductive system and breast disorders) | 0 | 6
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 5
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ferric Carboxymaltose (FCM) (N=996) | Standard Medical Care (SMC) (N=1022)
Constipation (Gastrointestinal disorders) | 9 | 79

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less